CLINICAL TRIAL: NCT03772197
Title: Head-to-Head Comparison of 18-Gene-Based Clinical-Genomic Model and Oncotype DX 21-Gene Assay for Predicting Recurrence of Early-stage Breast Cancer
Brief Title: Parallel Comparison of 18 Gene Classifiers and Oncotype DX (Nanostring)
Status: Completed | Type: Observational
Sponsor: Amwise Diagnostics Pte. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: RI-002
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Breast Cancer; Recurrence
Keywords: Breast cancer; Distant recurrence; NanoString; Gene-expression profiling; Prognosis; Locoreginal recurrence
MeSH Terms: conditions — Breast Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A recurrence index for distant recurrence (RI-DR), an 18-gene-based clinical-genomic model, has been developed for early-stage breast cancer (EBC). In this study, Investigators compared the prognostic performance of the RI-DR with the Oncotype DX (ODx) recurrence score (RS) for any recurrence risk type.

DETAILED DESCRIPTION:
With improved diagnosis, breast cancer can now be detected at early stages, thus improving survival rates. However, overtreatment is common; considering that the risk of recurrence is low, patients may suffer from side effects without receiving the full benefits of adjuvant therapies.

To overcome the imprecision of prognosis based on clinicopathologic factors, genomic tests for breast cancer prognosis, such as the Oncotype DX® (ODx), MammaPrint®, and EndoPredict® assay kits, are frequently utilized. These multigene panels were development based on Caucasian populations, and may not suitable to Asian population due to the differences in the incidence and lifestyle of breast cancer patients from different ethic backgrounds. To fiil this gap, an 18-gene classifier (18-GC) based on the gene-expression profiling of Chinese breast cancer patients was developed

In the current study, investigators combined clinical variables and genetic information to generate a clinical-genomic model: RI-DR, a recurrence index for distant recurrence (based on a genomic model and 6 clinical variables: age, tumor size, lymph node status, estrogen receptor status, lymphovascular invasion, tumor grading).

By using tissues that have been tested with ODx, in this study, investigators evaluated the performance of the RI-DR model with that of the ODx assay in the prognosis assessment of a cohort of patients from Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have performed (Oncotype Dx) genetic testing methods before June 30, 2017.
2. Surgery (mastectomy or breast preservation) as the first treatment.
3. ER or PR IHC positive
4. HER2 negative
5. N0-N1 patient
6. Available with FFPE tumor tissue

Exclusion Criteria:

1. T3-T4 or N2-N3
2. With distant metastasis before surgery
3. Preoperative chemotherapy / radiotherapy
4. Insufficient FFPE tumor samples

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: This study is a local validation and multi-center study. A total of 118 early-srage breast cancer (EBC) patients were included in this head-to-head comparison study, including 42, 15, and 81 patients treated between 2010 and 2016 at McKay Memorial Hospital, Koo Foundation Sun Yat-Sen Cancer Center, and National Taiwan University Hospital, respectively, in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
The locoregional recurrence (LRR) rate, within 5 years after surgery. | 5 years
  LRR risk calculated by 18-GC of breast cancer patients would be classified into high risk
The distant recurrence(DR) rate, within 5 years after surgery. | 5 years
  DR risk calculated by 18-GC of breast cancer patients would be classified into high risk

CONTACTS AND LOCATIONS:
Overall Officials: Skye Cheng, Principal Investigator — AMWISE DIAGNOSTICS PTE. LDT.
Locations (1):
- Amwise, Taipei, Taiwan